CLINICAL TRIAL: NCT03159390
Title: Human Metabolism of Ornithine Phenylacetate: A Study in Healthy Volunteers
Brief Title: Metabolism of Ornithine Phenylacetate
Acronym: OCERA OP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Ocera Therapeutics (Industry)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-0801
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: dietary supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- phenylacetate salt of ornithine (Experimental): There are 4 study days of approximately 10 hours. Amino acid tracers (e.g., OP, PHE, TYR) will be provided via IV. The dosage of OP provided in this study 6 g in a period of 6 hours. 2 muscle biopsies will be completed on 2 of the study days.
  Interventions: Other: phenylacetate salt of ornithine

INTERVENTIONS:
Other: phenylacetate salt of ornithine

SUMMARY:
Intravenous infusion of stable tracers of ornithine, glutamine, glutamate, and glycine will be performed, and collect blood samples, urine samples, and muscle biopsies to evaluate the effect of a continuous oral intake of phenylacetate salt of ornithine (OP) on its metabolic fate.

DETAILED DESCRIPTION:
The study involves 1 screening visit of approximately 1 hour and 4 study days of approximately 10 hours. The subject will be asked to arrive in the fasted state on all study days. Fasting prior to screening is not required. On the screening day, body weight and height will be measured and Dual-energy X-ray absorptiometry (DXA) will be performed to measure body composition. After 4 hours subjects received a continuous intravenous infusion with OP in a dosage of 1 g /h. Next to the stable tracers provided to determine OP metabolism, stable tracers of phenylalanine (PHE) and tyrosine (TYR) may be provided to determine the effect of OP on protein metabolism at plasma and muscle tissue level. This required 2 muscle biopsies and on 2 study days 1 set of stable tracer pulses.

ELIGIBILITY:
Inclusion criteria healthy subjects:

* Healthy male & female according to the investigator's or appointed staff's judgment
* Age 40-70 years (to be comparable with patients with liver cirrhosis: average 54.1 +/- 9.4 years)

Exclusion Criteria

* Metabolic diseases including diabetes and hepatic or renal disorders
* Presence of acute illness or metabolically unstable chronic illness
* Failure to give informed consent
* (Possible) pregnancy
* Any other condition according to the PI or nurse that would interfere with the study or safety of the patient or influence the results
* Unwilling to stop taking nutritional protein supplements within 5 days before test day
* History of hypo- or hyper-coagulation disorders, including use of a Coumadin derivative, history of deep venous thrombosis (DVT), or pulmonary embolism (PE) at any point in lifetime
* Currently taking anti-thrombotics (i.e. medical indication) and cannot stop for 3-7 days prior to test days
* Allergy to local anesthetic

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

PRIMARY OUTCOMES:
metabolism of ornithine phenylacetate to glutamate and glutamine | 4 study days that are 8 hours each
  The incorporation of the N atoms of ORN into glutamate, and the quantitative contribution of both pathways will be traced, and when the enrichment of ORN and GLU is measured in muscle tissue, give an estimation of the importance of muscle OAT for this incorporation.

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No